CLINICAL TRIAL: NCT01044212
Title: Bowel Function After Minimally Invasive Urogynecologic Surgery: A Prospective Randomized Controlled Trial
Brief Title: Bowel Function After Minimally Invasive Urogynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Gunhilde Buchsbaum, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29359
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Functional Disorder of Intestine
Keywords: Urogynecology
MeSH Terms: interventions — Dioctyl Sulfosuccinic Acid; Psyllium; Polyethylene Glycols; Bisacodyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docusate (Active Comparator): Docusate is the standard of care regimen
  Interventions: Drug: Docusate
- Bowel medications (Experimental): Docusate, Miralax, Metamucil wafers, Bisacodyl suppository
  Interventions: Drug: Bowel medications

INTERVENTIONS:
Drug: Docusate — Docusate 100mg BID
  Other Names: Colace
  Arms: Docusate
Drug: Bowel medications — Docusate 100mg BID Metamucil fiber wafers - 2 wafers daily Miralax 1 packet daily Bisacodyl 1 suppository BID
  Other Names: Colace; Psyllium; Polyethylene glycol; Dulcolax
  Arms: Bowel medications

SUMMARY:
The purpose of this study is to assess the effect of a standardized postoperative bowel regimen of over-the-counter medications in subjects undergoing minimally invasive urogynecologic surgery.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Planning to be admitted to the hospital to undergo minimally-invasive urogynecologic surgery at Strong Memorial Hospital.

Procedures may include:

* robot-assisted laparoscopic sacrocolpopexy
* sacrospinous ligament suspension
* uterosacral ligament suspension/paravaginal defect repair
* colpocleisis
* cystocele repair

Additional procedures may include:

* hysterectomy
* adnexectomy
* culdoplasty
* minimally invasive sling procedure (TVT or TOT)
* periurethral collagen injections
* enterocele repair

Exclusion Criteria:

* Planning to undergo laparotomy.
* Undergoing rectocele or perineocele repair as part of surgery.
* Taking Miralax, laxatives, enemas, or suppositories daily, at the time of enrollment.
* Presence of a colostomy.
* Chronic kidney disease
* Insulin-dependent diabetes mellitus
* Known cardiac disease
* Gastric ulcers
* Difficulty swallowing or esophageal stricture
* Persistent nausea and vomiting
* Signs and symptoms consistent with bowel obstruction

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunhilde Buchsbaum, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Candidates meeting criteria were offered participation at their preoperative visit.
Groups:
- Bowel Medications: Docusate, Miralax, Metamucil wafers, Bisacodyl suppository
  Bowel medications : Docusate 100mg BID Metamucil fiber wafers - 2 wafers daily Miralax 1 packet daily Bisacodyl 1 suppository BID
- Docusate Controls: Docusate is the standard of care regimen
  Docusate sodium : Docusate 100mg BID
Period: Overall Study
Arm/Group | Bowel Medications | Docusate Controls
Started | 35 | 37
Completed | 30 | 30
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bowel Medications | Docusate Controls | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 29 | 48
  >=65 years | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10) | 63 (9) | 61 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 37 | 72

OUTCOME MEASURES:

1. Primary Outcome: Time to First Post-op Bowel Movement
Description: The time to first post-operative bowel movement was measured in hours after surgery.
Time Frame: Within 1 week of surgery
Population: Power analysis
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bowel Medications | Docusate Controls
Number analyzed (Participants) | 30 | 30
hours | 64 (21) | 77 (24)

2. Secondary Outcome: Pain Level Associated With First Postoperative Bowel Movement
Description: The pain level experienced with the first post-operative bowel movement was recorded and measured on visual analog score with range 0 to 10 in units on scale. 0 being no pain at all. 10 being worst pain.
Time Frame: Within 1 week of surgery
Measure: Mean (Standard Deviation); unit: VAS pain score
Arm/Group | Bowel Medications | Docusate Controls
Number analyzed (Participants) | 35 | 37
VAS pain score | 3.6 (3.2) | 3.7 (2.8)

3. Secondary Outcome: Consistency of First Postoperative Bowel Movement
Description: The consistency of the first post-operative bowel movement was rated using the Bristol Stool Scale. This is a validated scale that is widely used. It is given to patients as a chart. The chart can be seen here: http://en.wikipedia.org/wiki/Bristol_stool_scale.
  The seven types of stool are:
  Type 1: Separate hard lumps, like nuts (hard to pass) Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft Type 5: Soft blobs with clear cut edges (passed easily) Type 6: Fluffy pieces with ragged edges, a mushy stool Type 7: Watery, no solid pieces. Entirely liquid
Time Frame: Within 1 week of surgery
Measure: Mean (Standard Deviation); unit: Bristol Stool Scale
Arm/Group | Bowel Medications | Docusate Controls
Number analyzed (Participants) | 35 | 37
Bristol Stool Scale | 3.13 (1.22) | 3.40 (1.07)

ADVERSE EVENTS:
Arm/Group | Bowel Medications | Docusate Controls
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37
Other Adverse Events (participants affected / at risk) | 0/35 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes